CLINICAL TRIAL: NCT05605925
Title: Ivermectin-artemisinin Combination Therapy for Eradication of Malaria
Acronym: IVIME
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Responsible Party: Principal Investigator, Dr. Mukonzo Jackson, Associate professor, Makerere University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MAKSHSREC-2021-237
Record Dates: First submitted 2022-02-17; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination; Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Active Comparator): 4 tabs artemether/lumefantrine 20/120mg, twice daily for 3 days
  Interventions: Drug: Artemether/lumefantrine
- Intervention arm (Experimental): IVN 600 mcg/kg/day for 3 days + 4 tabs artemether/lumefantrine 20/120mg, twice daily for 3 days
  Interventions: Drug: Artemether/lumefantrine; Drug: Ivermectin

INTERVENTIONS:
Drug: Artemether/lumefantrine — 4 tabs artemether/lumefantrine 20/120mg, twice daily for 3 days
Drug: Ivermectin — IVN 600 mcg/kg/day for 3 days
  Arms: Intervention arm

SUMMARY:
Malaria remains a leading cause of morbidity and mortality globally. Uganda has the 3rd highest global burden of malaria cases (5%) and the 7th highest level of deaths (3%), accounting for over 10,500 deaths annually. Uganda also has the highest proportion of malaria cases in East and Southern Africa (23.7%). Even with the current prevention strategies including use of impregnated mosquito nets, in 2017, malaria still accounted for 27-34 % of outpatient visits, 19-30 % of hospital admissions, up to 20% of all hospital deaths nationally. A significant percentage of deaths occur at home and are not reported by the facility-based Health Management Information System (HMIS). 27.2% of inpatient deaths among children under five years of age are due to malaria. The transmission of Plasmodium from humans to mosquitoes depends on the presence of mature gametocytes transmission stages. The current first-line treatment for uncomplicated falciparum malaria is artemether lumefantrine, an artemisinin combination therapy (ACT) which rapidly clears asexual parasites and developing gametocytes but leaves mature P. falciparum gametocytes largely unaffected, thus a proportion of patients may transmit malaria after successful ACT treatment and there is an urgent need to prevent this malaria transmission.

DETAILED DESCRIPTION:
Malaria remains a leading cause of morbidity and mortality globally, responsible for about one million deaths annually. 90% of these deaths occur in Africa, majority (90%) of whom are children under 5 years old, thus the focus of a global eradication campaign announced in 2007. Uganda has the 3rd highest global burden of malaria cases (5%) and the 7th highest level of deaths (3%), accounting for over 10,500 deaths annually. Uganda also has the highest proportion of malaria cases in East and Southern Africa (23.7%). Even with the current prevention strategies including use of impregnated mosquito nets, in 2017, malaria still accounted for 27-34 % of outpatient visits, 19-30 % of hospital admissions, up to 20% of all hospital deaths nationally. A significant percentage of deaths occur at home and are not reported by the facility-based Health Management Information System (HMIS). 27.2% of inpatient deaths among children under five years of age are due to malaria. Malaria has an indirect impact on the economy and development in general with socio-economic impact like out-of-pocket expenditure for consultation fees, drugs, transport to distant health facilities, such costs estimated to be as high as USD 3.88 per person per month (26 per household) or 3% of their annual income. Household expenditure for malaria treatment is also a high burden to the Ugandan population, consuming a larger proportion of the incomes in the poorest households. Additionally, malaria has a significant negative impact on the economy of Uganda due to loss of workdays because of sickness, decreased productivity, and decreased school attendance. Workers suffering from malaria may not be able to work for an estimated 5-20 days per episode and given that many people are at times infected multiple times a year, this has substantial financial consequences to families. Industries and agriculture also suffer due to loss of person-hours and decreased worker productivity and investors are usually wary of investing in such countries where malaria rates are high, leading to a loss in investment opportunities. Further, severe malaria impairs children's learning and cognitive ability by as much as 60%, consequently affecting the performance of Uganda's education programs. The transmission of Plasmodium from humans to mosquitoes depends on the presence of mature gametocytes transmission stages. The current first-line treatment for uncomplicated falciparum malaria is artemether lumefantrine, an artemisinin combination therapy (ACT) which rapidly clears asexual parasites and developing gametocytes but leaves mature P. falciparum gametocytes largely unaffected, thus a proportion of patients may transmit malaria after successful ACT treatment and there is an urgent need to prevent this malaria transmission. The current malaria prevention strategies in Uganda focus on the "keep healthy by avoiding malaria" phenomenon without the involvement of the host. Although key in malaria prevention, chemotherapeutic malaria preventive strategies are rarely used in Uganda since the currently available malaria prophylactic agents like mefloquine are only recommended for persons with short stay in malaria endemic settings. In short, to date there are limited malaria chemoprophylaxis options for resident Ugandans generally limiting the practice of malaria prevention.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with a laboratory malaria diagnosis who consent to participate in the study will be included.
2. Willingness to comply with all study procedures.
3. Adults patients aged 18-65 years.

Exclusion Criteria:

1. Participants with known hypersensitivity to Ivermectin
2. Patients with a history of asthma
3. Participants who live in a household of three or fewer people
4. Participants who reside more than 30km from the health care facility and have other members with suspected or confirmed malaria disease in their household at the time of enrolment.
5. Co-treatment with either strong cytochrome p-450 inducers including: rifampicin, carbamazepine and barbiturates or inhibitors: isoniazid, clofazimine that might potentially affect ivermectin disposition and clinical outcomes.
6. Loa loa as assessed by travel history to Angola, Cameroon, Chad, Central African Republic, Congo, DR Congo, Equatorial Guinea, Ethiopia, Gabon, Nigeria and Sudan in the last 4 years.
7. Active participation in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Malaria transmission rates in a household | Malaria Transmissibility from index participant to other household members within 28 days
  Malaria transmission rates in a household from an index participant. Index participant is participant who is first diagonised with malaria in that household. The transmission will be assessed using nanopore sequencing to assess for similarity between the malaria falciparum agent of the index participant and that of an household member

SECONDARY OUTCOMES:
Safety of ivermectin-artemether/lumefantrine in malaria infected patients | daily for 30 days while following up participant
  Safety of the the use of ivermectin-artemether/lumefantrine in malaria infected patients shall be assessed using the adverse events score scale of 1-mild, 2-moderate, 3-severe, 4-life threatening and 5-death

CONTACTS AND LOCATIONS:
Locations (1):
- ST. Paul's Health Center, Kasese, Uganda

IPD SHARING:
Plan to Share IPD: No